CLINICAL TRIAL: NCT03783351
Title: CYP2C19 Genotype-GUided Dual Antiplatelet theRapy in pAtieNts Treated With New Generation Drug Eluting stEnts (the GUARANTEE Study)
Brief Title: Genotyping GUided Antiplatelet theRapy in pAtieNts Treated With Drug Eluting stEnts (GUARANTEE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUARANTEE
Record Dates: First submitted 2018-12-11; First posted 2018-12-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Angina, Stable; Acute Coronary Syndrome; Drug-Eluting Stents; Genotype
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (No Intervention): Patients randomized to the Conventional Therapy arm will receive either clopidogrel or ticagrelor, according to the clinical and procedural characteristics of patients. CYP2C19 genotyping will be performed at the end of study.
- CYP2C19 Genotyping (Active Comparator): CYP2C19 genotyping will be performed within 48 hours after randomization. CYP2C19 *2 or *3 reduced function allele patients will receive ticagrelor 90 mg bid, whereas non-*2 or -*3 CYP2C19 patients will receive clopidogrel 75 mg once daily.
  Interventions: Genetic: CYP2C19 genotype testing

INTERVENTIONS:
Genetic: CYP2C19 genotype testing — CYP2C19 genotype testing will be conducted in a designated central laboratory.
  Other Names: clopidogrel; ticagrelor
  Arms: CYP2C19 Genotyping

SUMMARY:
The aim of this study is to assess the efficacy and safety of the CYP2C19 genotype guided antiplatelet treatment strategy, using clopidogrel in non-carriers of a CYP2C19*2 or *3 allele and ticagrelor in carriers of a CYP2C19*2 or *3 allele in patients treated with new generation drug eluting stents.

DETAILED DESCRIPTION:
Background: P2Y12 receptor inhibitors are crucial for the management of patients undergoing coronary stenting. Although large-scale trials have shown that ticagrelor is superior to clopidogrel in terms of platelet inhibition and reduction of major adverse cardiovascular events (MACE), clopidogrel remains the most commonly used P2Y12 receptor inhibitor due to its lower price and bleeding risk. Despite the combined use of aspirin and clopidogrel, a substantial portion of patients after coronary stenting are at increased risk for adverse cardiovascular events including death, myocardial infarction, and stent thrombosis. This phenomenon may be due to the so-called clopidogrel resistance. Cytochrome P450 2C19 (CYP2C19) polymorphism plays a crucial role in the clopidogrel resistance. CYP2C19 is responsible, in part, for converting the clopidogrel prodrug into an active metabolite that irreversibly binds to the P2Y12 receptor thus inhibiting ADP-induced platelet aggregation. CYP2C19*2 and *3, which encounter loss function, have been demonstrated to be the most common genetic variants resulting in clopidogrel resistance.

Methods: Patients who undergo coronary stenting will be randomized to a prospective CYP2C19 genotype-guided antiplatelet therapy arm versus a conventional therapy arm. Venous blood collection will be completed immediately after randomization in all patients eligible for the study. The genotype results involving CYP2C19*2 and *3 allele variants will be obtained within 48 hours only in the genotyping arm. CYP2C19 *2 or *3 reduced function allele patients will receive ticagrelor 90 mg bid, whereas non-*2 or -*3 CYP2C19 patients will receive clopidogrel 75 mg once daily. The conventional therapy arm will receive either clopidogrel or ticagrelor, according to the clinical and procedural characteristics of patients. The dual antiplatelet therapy will last for at least one year in the both arms. The primary endpoints will be evaluated at one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years of age
* Patient presents with acute coronary syndrome (ACS) or stable coronary artery disease (SCAD)
* Patient has a percutaneous coronary intervention (PCI) indication and the new generation drug eluting stent(s) is successfully implanted

Exclusion Criteria:

* Patient unable to receive 12 months of dual anti-platelet therapy
* Patient developing procedure-related complications such as stent thrombosis, coronary dissection, coronary perforation, cardiac tamponade or no-reflow during PCI
* Contraindicated or allergic to clopidogrel or ticagrelor
* Patient or physician refusal to enroll in the study
* Patient having received thrombolytic therapy within the previous 24 hours
* Physician has known the patient's CYP2C19 genotype
* Anticipated discontinuation of dual anti-platelet therapy within the 12-month follow-up period, example for elective surgery
* History of intracranial hemorrhage
* Patient has a history of bleeding diathesis or coagulopathy
* Patient has an active pathological bleeding, such as active gastrointestinal (GI) bleeding
* Patient is pregnant, breastfeeding, or planning to become pregnant within 12 months
* Patient is receiving chronic oral anticoagulation therapy (i.e., vitamin K antagonist, direct thrombin inhibitor, Factor Xa inhibitor)
* Patient with cardiogenic shock or mechanical circulatory assist devices placed
* Patient with LVEF <30%
* Patient with active liver diseases
* Patient with severe renal insufficiency (eGFR <30ml/min/1.73m2 based on simplified MDRD equation or CrCl <30ml/min based on Cockcroft-Gault equation)
* Patient has a malignancy or a life expectancy of less than one year
* Platelet count <100 000/μL, or hematocrit <32% or >52%, or white blood cell count <3000/μL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4009 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of main adverse cardiovascular and cerebrovascular events (MACCE) | 1 year
  MACCE will include all-cause death, non-fatal stroke, non-fatal myocardial infarction (MI) and ischemia driven revascularization at one-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, PhD,MD, Study Chair — Beijing Anzhen Hospital; Xiaoli Liu, PhD, MD, Study Director — Beijing Anzhen Hospital; Xiaoteng Ma, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (9):
- China (9):
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Tong Ren Hospital, Beijing, Beijing Municipality
  - Beijing LuHe Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No